CLINICAL TRIAL: NCT04926987
Title: The Research of Human Cortex Cell Atlas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-030
Record Dates: First submitted 2021-05-29; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Aging; Epilepsy; Trauma, Brain
Keywords: Single-Cell Analysis; aging; epilepsy; trauma brain
MeSH Terms: conditions — Epilepsy; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tissue

INTERVENTIONS:
Other: brain tissue single-cell sequencing — Using single-cell sequencing to study the brain tissue single-cell transcriptome difference in aging, epilepsy, and mental disorders

SUMMARY:
In this study, the single-cell transcriptome sequencing technology was used to study the transcriptome differences at the single-cell level in normal human brain, aging human brain, and epileptic brain.

DETAILED DESCRIPTION:
The human brain has about 100 billion cells and makes up neural networks.The abnormal activity of neurons can affect the operation of neural networks, leading to neurological diseases.With the coming of the age of global population aging, neurodegenerative diseases such as Alzheimer's, Parkinson's and Huntington's have become an increasing burden on human health.

Cells are the basic unit of brain. Understanding the mechanism of brain activities includes not only the mechanism of neural network, but also the self-regulation of its basic unit, that is, the regulation of gene expression based on brain activity.The abnormal expression and regulation of genes lead to the abnormal activities of the nervous system.Therefore, studying the regulation mechanism of gene expression at the cellular level is an important way to research brain diseases.The recent development of single-cell RNA-sequencing technology provides a possibility to understand the functioning mechanism of the brain at the cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Craniocerebral injury patients needing operative treatment
* Treatment-resistant epilepsy patients needing resection surgery

Exclusion Criteria:

* Vital signs unstable
* Pregnancy
* Tumor
* Incomplete medical history, imaging and clinical diagnosis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Craniocerebral injury patients needing operative treatment
  2. Treatment-resistant epilepsy patients needing resection surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
single-cell RNA sequencing | 1 Day of surgery
  single-cell RNA sequencing resultes of brain sample

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Zhang, M.D, Study Chair — Department of Neurosurgery; Junming Zhu, M.D, Principal Investigator — Department of Neurosurgery
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China